CLINICAL TRIAL: NCT03897504
Title: Surgical Evaluation Of Using The Inner Surface Of The Prepuce In Feminizing Genitoplasty In Cases Of Verilized Females With Congenital Adrenal Hyperplasia
Brief Title: Surgical Evaluation of Using the Prepuce in Feminizing Genitoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Tarek Mohamed Bahget, Assistant lecturer, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-100-2018
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: congenital adrenal hyperplasia; Feminizing genitoplasty; Vaginal stenosis
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- feminizing genitoplasty using inner surface of the prepuce (Experimental): Feminizing genitoplasty will be done using the prepuce as a pedicled tubularized flap to create the new vagina, the new vagina which the investigators create it from the prepuce will be sutured above to the native vagina after its separation from the urogenital sinus, and the remaining part of the urogenital sinus will be used to create the urethra, the remaining part of the prepuce will create the labia minora, clitoroplasty will be attempted in all patients.
  Interventions: Procedure: feminizing genitoplasty using inner surface of the prepuce as pedicled tubularized flap

INTERVENTIONS:
Procedure: feminizing genitoplasty using inner surface of the prepuce as pedicled tubularized flap — the prepuce of the females with congenital adrenal hyperplasia will be tubularized and used as pedicled flap in creating the new vagina, the urethra will be completed with the urogenital sinus, no mobilization either partial or complete urogenital mobilization will be needed in cases with low and intermediate confluence level (less than 30 mm), in case with high confluence (more than 30 mm) laparoscopic vaginal pullthrough will be attempted first then the same previously described technique will be applied, the depth of the confluence will be determined before starting surgery by doing genitograph under general anaesthesia, stent will be kept in the new vagina for 5 days and further scheduled calibrations and dilatations will be applied regularly with paying attention to urinary complications like incontinence and urethrovaginal fistula by doing urodynamics and micturating cystourethrogram if there is a complain.

SUMMARY:
Background and Rationale: The vaginoplasty remains a challenge for the surgeon. The most commonly used techniques have been: the Y-V plasty described by fortunoff for low vagina, the pullthrough operation described by Hendren and Crawford for high vagina, and the passerini-Glazer technique . None of these procedures is entirely satisfactory; with the first two, the neovagina has a tendency to become stenotic in most cases. Moreover, in the third, in addition to the high rate of stenosis, which is encountered in a third of case , the high rate of urethro-vaginal fistulas is unacceptable

Objectives :

To describe and evaluate a surgical technique for vaginoplasty that is easy to realize with fewer complications especially vaginal stenosis.

Study population & Sample size : 24 patients suffering from congenital adrenal hyperplasia (CAH) presenting to outpatient clinic of diabetis Endocrine And Metabolism Pediatric Unit (DEMPU) of Cairo University Specialized Pediatric Hospital will be considered.

Study Design : non-controlled prospective clinical trial with all patients included in single group

Methods: Cystoscopy will be done promptly before proceeding to surgery, Confluence depth more than 20 mm is considered high anomaly, feminizing genitoplasty will be done as a one-stage procedure, One month after operation, examination under anesthesia will be done with calibration of vagina.

Possible Risk (s) to study population : The risk of this study is involving a vulnerable group of females which exposed to lengthy operation may complicate with bleeding and need for blood transfusion, infection early after surgery or vaginal stenosis.

Outcome parameter (s):

Vaginal calibration using hegars dilators Urodynamics for females older than 3 years and complaining from incontinence

DETAILED DESCRIPTION:
• Background and Rationale: Disorders of sex development(DSD) are medical conditions in which the development of chromosomal, gonadal, or anatomic sex varies from normal and may be incongruent with each other. Five main groups of DSD patients may be identified, submitted to the gender assignment process, and may be considered for a surgical genital reconstruction. (Lee Pa et al, 2006) Congenital adrenal hyperplasia (CAH) refers to a group of autosomal recessive disorders resulting from deficiency of one of the five enzymes required for synthesis of cortisol in the adrenal cortex. CAH is the most common cause of genital ambiguity. (van der Zwan, 2013) About 90-95% of individuals with CAH have a mutation in CYP21A2 gene, encoding 21-hydroxylase enzyme. The worldwide incidence of classical 21 OHD is 1:15,000 to 1:16,000 live births of which approximately 75% are salt wasters. That leads to a block of normal production of cortisone and results in overproduction of steroid metabolism by-products through pituitary feedback. These androgenic steroids lead to a variable degree of masculinization of normal female fetus.

The goal of therapy in CAH is to both correct the deficiency in cortisol secretion and suppresses adrenocorticotropic hormone (ACTH) overproduction. Proper treatment with glucocorticoid reduces stimulation of the androgen pathway, thus preventing further virilization and allowing normal growth and development. In addition to hormonal therapy, feminizing reconstructive surgery targets the correction of anatomical disturbance. The feminizing genitoplasty operation consists of reducing the size of the phallus (clitoroplasty), creating labia minora and vaginoplasty.

• Sample size: Sample size calculation: n = 2(Za+Z1-β)2σ2/Δ2 n sample size Za = 1.65 ( p<0.05 as acceptable and a study with 80% power; using the below table, we get the following values: Zα, is 1.65 a error 5% 1% .1% 2 sided 1.96 2.5758 3.2905

1 sided 1.65 2.33 Z1-,β= 0.8416 power 80% 85% 90% 95% value 0.8416 1.0364 1.2816 1.6449 σ standard deviation =0 .5 Δ effect size 36% =0.36 Effect of using the prepuce in minimizing vaginal stenosis is 100% - effect of using other techniques 64%

N =2(1.65+0.8416)2 0.52 / 0.362 = 24 patients.

• Study Design: non-controlled prospective clinical trial with all patients included in single group.

* Ethical committee approval : approved (N-100-2018)
* Study Methods

Population of study & disease condition:

24 patients suffering from congenital adrenal hyperplasia (CAH) presenting with virilized external genitalia to outpatient clinic of diabetes Endocrine And Metabolism Pediatric Unit (DEMPU) of Cairo University Specialized Pediatric Hospital will be considered.

Methodology in details :

Patient recruitment females with congenital adrenal hyperplasia presenting with persistent urogenital sinus and virilized external genitalia to the outpatient clinic of Diabetes Endocrine And Metabolism Pediatric Unit (DEMPU) of Cairo University Specialized Pediatric Hospital

Pre-operative management History taking laying stress on age at diagnosis, family history of similar conditions and consanguinity in addition to any salt losing events.

Reviewing the patients charts for the investigations (basal adrenal precursors, karyotype, pelvic ultrasound) Complete genital examination to detect the degree of virilization (number and types of openings, the presence of rugae or pigmentation, phallus size and Prader scale).

Routine pre-operative blood tests will be done .

Perioperative hormonal therapy in the form of hydrocortisone and/or fludrocortisone in conjunction with pediatric anesthesia and pediatric endocrinology teams including dose adjustment and electrolytes follow up.

Genitography: Patient is generally anesthetized either in same setting of surgery or pre-operatively in different setting, The depth of confluence from perineal marker is measured in ratio to perineal marker dimensions whatever the scale of genitography picture is, then measurements are taken in millimeters. Other measurements of proximal urethra and vagina to the confluence are taken.

Operative technique Cystoscopy will be done promptly before proceeding to surgery in the same setting.

Confluence depth more than 20 mm is considered high anomaly with consequent difficult and lengthy procedure with high probability of need to use vaginal pullthrough in combination with the use of inner layer of the prepuce.

feminizing genitoplasty will be done as a one-stage procedure. The patient is placed in the lithotomy position for the best exposure of the perineum. A Foley catheter French 6 is placed in the vagina to facilitate identification of structures during dissection, The clitoroplasty will be attempted in all Cases.

The dissection of the flap from the inner surface of the prepuce with its pedicle will be done after measuring the distance between the native vagina and perineum. and then tubularized onto a rectal stent (French 12 or 14).

The proximal edge of the preputial flap will be sutured to upper vagina and its distal edge to outer edge. The rectal drain will be left in the vagina for 5 days postoperatively, by this technique the vaginoplasty can be achieved without further mobilization of the vagina which may affect the continence of the patient if we divide pubourethral ligament, labia this procedure will be followed by clitoroplasty and labioplasty.

In cases of low urogenital sinus (less than 2 cm), the use of preputial flap alone is often sufficient.

in case of high confluence additional procedure will be done in the form of laparoscopic vaginal pull-through

Postoperative management:

Wound will be closed by x-shaped bandage for 24 hours.

Vitamin K, ethamsylate (dicynone) and tranexamic acid (cyklokapron) will be given to help in hemostasis.

After dressing removal the wound will be left exposed and flushed with sterile -saline every 4-6 hours

Urinary catheter and vaginal stent will be removed on 5th to 7th day post operatively.

Parenteral broad spectrum antibiotics and antianaerobes will be given for one week. Stress doses of steroids will be continued for 2-3 days after surgery at double usual oral dose followed by tapering and returning to the original dose

postoperative management: One month after operation, examination under anaesthesia will be done with calibration of vagina using Hegar dilators and making decision for further need for repeated vaginal dilatation.

Urodynamics will be applied for patients older than 3 years old to asses the continence in cases with high confluence.

Primary outcome:

To calibrate the vagina and asses the degree of vaginal stenosis if present and need for further vaginal dilatation.

Secondary outcome:

To asses other outcomes specially the continence in patients older than 3 years old and the prescence of urethrovaginal fistula.

Short term complications:

* Infection at vestibule and incision lines
* accidental removal of the catheter
* haematoma
* secondary haemorrage

Intermediate and long term complications:

* urethrovaginal fistula
* recurrent persistant urogenital sinus (UGS)
* Vaginal stenosis
* Urinary incontinence

ELIGIBILITY:
Inclusion criteria:

* Females (46, XX genotype identified by karyotype
* Age: infants and children from 18 months old age to 14 years
* Virilized external genitalia.
* Persistent urogenital sinus
* Congenital adrenal hyperplasia.
* Controlled by glucocorticoid and mineralocorticoid replacement therapy and clinically and hormonally judged fit for surgical interventions.
* Voluntarily provided informed written consent of the parents for the planned procedure and possible risks.
* Informed written approval of the parents of the included children to use clinical data collected in a research program.

Exclusion Criteria:

* Male disorders of sexual development (46 XY)
* Debatable sex of rearing; Mixed gonadal dysgenesis, Ovotesticular disorders of sexual development and partial androgen insensitivity syndrome.
* Inadequate compliance with corticosteroid therapy, rendering surgery or interventions clinically hazardous or unsuitable.
* Inadequately controlled hormonal assay: elevated androgens.
* Patients who did any corrective surgery before.

Ages: 18 Months to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — the study applicable only in over virilized females with congenital adrenal hyperplasia
Enrollment: 5 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
vaginal size calibration | 6 months to one year
  the new vagina will be assessed for stenosis 1 month after the procedure using Hegar dilators under general anaesthesia, further calibration will be done over 6 months to ensure patency of the vagina and to avoid stenosis by dilatation if stenosis encountered

SECONDARY OUTCOMES:
urinary incontinence | 6 months
  in patient older than 3 years and complaining from incontinence, urodynamics will be done.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine- Cairo University, Cairo, El Manial, Egypt